CLINICAL TRIAL: NCT00347529
Title: A Randomised Double Blind Dose-Ranging Study to Assess the Safety, Tolerability and Immunogenicity of a Monovalent H5 DNA Influenza Vaccine (A Vietnam/1194/2004) Administered by Particle Mediated Epidermal Delivery (PMED) to Healthy Adults
Brief Title: Safety Study of an Influenza Vaccine Against a Potential Pandemic Strain of Flu
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PowderMed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PM FLP-001
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2007-01

CONDITIONS: Influenza (Pandemic)
Keywords: DNA vaccine, influenza, immunogenicity, tolerability, PMED, pandemic
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: pPML7789 with and without pPJV2012 administered by PMED

SUMMARY:
The purpose of this study is to evaluate how well the vaccine is tolerated at sites where administrations are given, any effects it may have on subjects' wellbeing and whether it can produce antibody responses in the body that may protect against the subjects catching a pandemic strain of flu

DETAILED DESCRIPTION:
Pandemic influenza occurs when a strain of influenza to which the human population has not been exposed develops the ability to infect man and spread from person to person. Some pandemics can have very severe health impacts and be widespread. This study will evaluate PowderMed's Particle Mediated Epidermal Delivery (PMED) DNA vaccine for pandemic influenza as a potential alternative to other vaccine technologies. This study represents the first study with this vaccine and will provisionally assess its safety and immunogenicity (ability to generate an immune response) at four different dose combinations. The vaccine will be given as a prime-boost regimen with vaccination on Days 0 and 28

ELIGIBILITY:
Inclusion Criteria:

Healthy adults volunteers (women must be of nonchild-bearing potential) Provided written informed consent

-

Exclusion Criteria:

No significant concomitant illness No allergy to gold No immunosuppression due to disease or treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75
Dates: Start 2006-08; Study Completion 2007-01

PRIMARY OUTCOMES:
Safety, tolerability and local reactogenicity-AEs and laboratory parameters.

SECONDARY OUTCOMES:
Immunogenicity of the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Tim Mant, BSc, FRCP, FFPM, Principal Investigator — Guys Research Drug Unit, Quintiles UK Ltd.
Locations (1):
- Guys Research Drug Unit, Quintiles Ltd., London, United Kingdom